CLINICAL TRIAL: NCT06741488
Title: Adherence of Women With Fibromyalgia to Home Exercise Programme and Perceived Barriers to Exercise
Brief Title: Fibromyalgia, Exercise Adherence and Barriers
Status: Not yet recruiting | Type: Observational
Sponsor: Konya Beyhekim Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Savaş Karpuz, Associate Professor, Konya Beyhekim Training and Research Hospital
Other Study IDs: 2024-10-05
Record Dates: First submitted 2024-12-05; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- fibromyalgia: No intervention will be made. The questionnaire will assess adherence to exercise and perceived barriers.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — Exercise Adaptation Rating Scale

SUMMARY:
We aimed to investigate adherence to exercise and perceived barriers to exercise in patients with fibromyalgia who were advised to exercise.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with fibromyalgia according to ACR 2016 criteria
* Female
* To be informed about the benefits of exercise, the importance of exercise compliance and to be shown the exercise program in practice and to be given a printed form

Exclusion Criteria:

* Having a systemic or mental disease that may prevent exercise

Ages: 18 Years to 65 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — self-report
Study Population: physical medicine and rehabilitation outpatient clinic
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
exercise adherence | one month after the exercise is recommended
  Exercise Adaptation Rating Scale, Total score ranges from 0-64, with higher scores indicating greater adherence
perceived barriers to exercise | one month after the exercise is recommended
  Benefits/barriers to exercise scale, The score range of the barrier scale is 14-56 and the score range of the benefit scale is 29-116. The sum of all items in the scale gives the total score of the scale and a high total scale score indicates that the individual finds exercise useful.